CLINICAL TRIAL: NCT00964080
Title: A Phase Ib/II Study of MBP-426 in Patients With Second Line Gastric, Gastro Esophageal, or Esophageal Adenocarcinoma
Brief Title: Study of MBP-426 in Patients With Second Line Gastric, Gastroesophageal, or Esophageal Adenocarcinoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mebiopharm Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBP-426 201
Record Dates: First submitted 2009-08-17; First posted 2009-08-24 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2012-04

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study of MBP-426/leucovorin/5-FU (Experimental): Study of MBP-426/leucovorin/5-FU. MBP-426 will be administered at a dose of 170 mg/m2 every three weeks. Leucovorin will be administered ata dose of 400 mg/m2 after the MBP-426 infusion and in the absence of allergy/infusion reaction. 5-FU is administered concurrently with the leucovorin infusion and after the MBP-426 administration as a 46-hour continuous infusion of 2400 mg/m2.
  Interventions: Drug: MBP-426/Leucovorin/5-FU

INTERVENTIONS:
Drug: MBP-426/Leucovorin/5-FU — MBP-426 will be administered at a dose of 170 mg/m2 every three weeks. Leucovorin will be administered at a dose of 400 mg/m2 after the MBP-426 infusion and in the absence of allergy/infusion reaction. 5-FU is administered concurrently with the leucovorin infusion and after the MBP-426 administration as a 46-hour continuous infusion of 2400 mg/m2.
  Other Names: Liposomal Oxaliplatin/Folinic Acid/5-Fluorouracil

SUMMARY:
The ongoing study is a Phase II, open-label study to evaluate the efficacy of MBP-426 at a dose of 170 mg/m2 in combination therapy in patients with second line metastatic gastric, gastro-esophageal junction or esophageal adenocarcinoma.

DETAILED DESCRIPTION:
This study will start with a Phase Ib portion, at a dose of 226 mg/m2, a dose in which good tolerability was demonstrated in the Phase I trial. A cohort may be enrolled at 301 mg/m2, if 226 mg/m2 is well tolerated. The dose determined from the Phase Ib portion of the study will then be evaluated in the Phase II portion.

This design will permit evaluation of a true positive or negative response while limiting over exposure of patients to the study drug. If this regimen does offer a positive response, its reduced toxicity and potentially greater efficacy may yield better outcomes for patients requiring second-line therapy for UGI cancer.

Following completion of the Phase Ib part of the present trial, the dose recommended for use in the Phase II part is 170 mg/m2 MBP-426.

ELIGIBILITY:
Inclusion Criteria:

Phase Ib:

1. Advanced or metastatic solid tumor malignancy that is refractory to STD therapy, or that has relapsed after STD therapy, or for which conventional therapy is not reliably effective, or no effective therapy is available.
2. Measurable disease as defined by RECIST. If recurrence is documented following radiation therapy, the recurrence must have occurred outside the radiation field. Lesions which are located within a previously irradiated field are not considered measurable.
3. Age ≥18.
4. ECOG performance status: 0, 1 or 2.
5. Adequate organ and system function:

   * Bone marrow: ANC ≥1500/mm3, platelet count ≥100000/mm3, and Hb ≥9 g/dL;
   * Coagulation: PT <1.3 x ULN, PTT >LLN, <1.1 x ULN
   * Renal: Serum creatinine of ≤1.5 x the institution's ULN or calculated creatinine clearance ≥60 mL/min/1.73m2;
   * Hepatic: Total bilirubin ≤1.5 mg/dL, ALT and AST ≤2.5 x ULN (or 5 x ULN), and ALP ≤2.5 x ULN (or 5 x ULN).
6. Recovered to ≤Gr 1 from all acute toxicities caused by prior cancer therapies except for residual toxicities which do not pose an ongoing medical risk.
7. If of childbearing potential, agree to use an effective method of contraception prior to study entry, for the duration of the study, and for 30 days after the last dose of MBP-426 with FA/5-FU. A negative pregnancy test must be documented at baseline. Patients may not breastfeed while in this study.
8. Have the ability to maintain a central IV access.
9. Able to comply with the protocol treatments and procedures.
10. Provide written informed consent indicating that they are aware of the investigational nature of this study and in keeping with the institution's policies.

Phase II:

1. Inoperable, histologically, or cytologically confirmed, locally advanced or metastatic gastric, GE junction, or esophageal adenocarcinoma that has recurred or progressed following 1 prior chemotherapy.
2. Measurable disease as defined by RECIST. If recurrence is documented following radiation therapy, the recurrence must have occurred outside the radiation field. Lesions which are located within a previously irradiated field are not considered measurable.
3. ECOG performance status: 0 or 1.
4. Identical to criteria numbers 3-10 for Phase Ib portion of the study.

Exclusion Criteria (Phase Ib and II):

1. Major surgery within 14 days prior to study enrollment.
2. Radiotherapy, hormonal therapy, immunotherapy, or investigational agents within 30 days of enrollment (6 weeks for mitomycin C). A washout is required for chemotherapy, antibodies and small molecules, equivalent to at least 5 half-lives or 30 days, whichever is shorter, prior to study entry. Concurrent use of bisphosphonates is permitted.
3. Have had a past or have a current 2nd primary malignancy (except in situ carcinoma of the cervix or adequately treated nonmelanomatous carcinoma of the skin, or other malignancy treated at least 3 years previously with surgery and/or radiotherapy and no evidence of recurrence since that time).
4. Known or clinical evidence of CNS metastases.
5. Receiving high-dose steroids more than a dexamethasone-equivalent dose of 4 mg/day.
6. Current active infections requiring anti-infectious treatment.
7. Significant intercurrent illnesses that would have compromise the safety of the patient or compromise the ability of the patient to complete the study.
8. Documented or known hematologic malignancy and/or bleeding disorder.
9. Peripheral neuropathy ≥Gr 2 (NCI-CTCAE, Ver. 3.0).
10. Any requirement(s) for therapeutic anticoagulation that increases INR or aPTT above the normal range (low dose DVT or line prophylaxis is allowed).
11. Have NYHA Class 3 or 4 heart disease, active ischemia, or any uncontrolled, unstable cardiac condition for which treatment for the condition is indicated but is not controlled despite adequate therapy.
12. History of allergy to any of the treatment components (oxaliplatin, 5-FU, FA, liposome, ferritin).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-10 (Actual); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
To determine the dose of MBP-426 for use in the Phase II portion of this study of MBP-426 administered every 21 days in combination with leucovorin (folinic acid or FA) and fluorouracil (5-FU) | 4 months

SECONDARY OUTCOMES:
To characterize the safety profile of the combination therapy | 4 months
To determine the plasma and urine pharmacokinetics of MBP-426 when given in combination with leucovorin and 5-FU | 4 months
To undertake a preliminary exploration of anti-tumor activity of the combination therapy | 4 months
To characterize the safety profile of the combination therapy | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer A. Ajani, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (5):
- United States (3):
  - Mary Crowley Medical Research Center, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
- Georgia (2):
  - A.Gvamichava National Center of Cancer, Tbilisi
  - Medulla Chemotherapy and Immunotherapy Clinic, Tbilisi

REFERENCES:
- [Derived] Alavi N, Rezaei M, Maghami P, Fanipakdel A, Avan A. Nanocarrier System for Increasing the Therapeutic Efficacy of Oxaliplatin. Curr Cancer Drug Targets. 2022;22(5):361-372. doi: 10.2174/1568009622666220120115140. PMID 35048809